CLINICAL TRIAL: NCT05510479
Title: Post-market Study for At-home Evaluation of Near Visual Acuity With OdySight, a Smartphone Based Medical Application in Comparison to a Standardized Method (TIL002)
Brief Title: Post-market Evaluation of OdySight App to Monitor Near Visual Acuity at Home (TIL002)
Acronym: TIL002
Status: Completed | Type: Observational
Sponsor: Tilak Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-A03583-36
Record Dates: First submitted 2022-07-19; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Visual Impairment
Keywords: Visual acuity; Digital therapeutics; Medical software; ETDRS; Macular Edema; Age-related Macular Degeneration
MeSH Terms: conditions — Vision Disorders; Macular Edema; Macular Degeneration | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- OdySight vs Standardized methods: All patients perform Visual Acuity testing through OdySight and according to standard practice
  Interventions: Other: Software as medical device

INTERVENTIONS:
Other: Software as medical device — At home measurements of visual acuity through a mobile app

SUMMARY:
OdySight is a mobile application allowing self-testing of visual parameters including near visual acuity and communication of the data to an online dashboard to patient's doctors. TIL-002 post-market clinical trial objective is to evaluate the near visual acuity at home, measured with OdySight application in comparison to the standardized methods. The clinical trial is intended to prove that OdySight can provide relevant data and participate in the remote monitoring of subject vision.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria:

1. Age ≥ 18 years, all genders
2. Affiliated to or beneficiary of the French health care system
3. Signed/written informed consent
4. Already user of Odysight on a compatible smartphone/tablet
5. Patients willing and able to comply with all study and follow-up procedure

   Ophthalmic inclusion criterion:
6. Baseline binocular visual acuity with habitual correction ≥ 20/63 (3/10) AND with at least an eye ≥ 20/200 (1/10).

Exclusion Criteria:

General exclusion criteria:

1. Any pathology that is considered by the investigator as capable of affecting the quality of the main evaluation criteria.
2. Any planned surgery likely to modify patient refraction during the study (cataract surgery for example)
3. Subject not considered by the investigator or designee to correctly use ODYSIGHT modules
4. Subject unable to recognize alphabet letters or unable to correctly distinguish body laterality
5. Not French speaking patient
6. Epileptic users

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with a near visual acuity between 0.0 and 1.0 logMAR in at least one eye, and binocular VA equal to or better than 0.5 logMAR are targeted for this study.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Equivalence between OdySight and standardized methods - Near Visual Acuity | 2 months
  To assess the equivalence between a smartphone based evaluation of near visual acuity with ODYSIGHT at home and standardized methods (Sloan ETDRS near vision letter chart and Landolt C near vision chart) performed in clinic.

SECONDARY OUTCOMES:
Equivalence between OdySight and standardized methods - 4-meter distance Visual Acuity | 2 months
  ETDRS visual acuity at a 4-meter distance at clinic and near visual acuity evaluated with ODYSIGHT at home.

OTHER OUTCOMES:
Near Visual Acuity - Subgroups analysis | 2 months
  To assess the equivalence between a smartphone based evaluation of near visual acuity with ODYSIGHT at home and with standardized methods in specific subgroups defined by visual acuity and by pathology
Near Visual Acuity variability | 2 months
  To assess variability of measurements with a smartphone-based evaluation of NVA with Odysight at home vs at clinic
Vision changes tracking | 2 months
  To evaluate ability of the VA application module to track vision change over time as compared to standardized methods.
Compliance to OdySight | 2 months
  To evaluate compliance of daily use among time.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Ophtalmologique Rabelais, Lyon
  - Institut Ophtalmologique de l'Ouest Clinique Jules Verne, Nantes
  - Centre Hospitalier National d'Ophtahlomogie du Quinze-Vingts, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No